CLINICAL TRIAL: NCT02307604
Title: Screening Platform of EORTC for Clinical Trials Access in Brain Tumors
Brief Title: SPECTAbrain: Screening Patients With Brain Tumors for Efficient Clinical Trial Access
Acronym: SPECTAbrain
Status: Withdrawn | Type: Observational
Why Stopped: This study has been merged with 1553 SPECTA, in which brain patients are enrolled
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1313
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Brain Neoplasms
Keywords: Brain tumor; Biomarkers; Screening
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — FFPE blocks of tumour tissue Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Brain cancer: Patients with diagnosis of brain cancer at any stage
  Interventions: Genetic: Tumour markers testing

INTERVENTIONS:
Genetic: Tumour markers testing

SUMMARY:
The SPECTAbrain protocol describes a structure for screening patients with brain tumors to efficiently allocate eligible patients in relevant therapeutic biomarker-driven clinical trials. Efficiency is promoted through the creation of a clinical database of brain tumor patients and the respective human biological material biobank for molecular characterization. The main objectives are to:

* Allocate patients to clinical trials according to the clinical characteristics and molecular profile of their tumor;
* Identify or validate new molecularly defined subgroups of tumors;
* Investigate the prevalence of novel biomarkers to plan future clinical trials;
* Enable exploratory/future research;
* Facilitate establishment of quality-assured and validated tests for Central Nervous System (CNS) tumor biomarkers;

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed newly diagnosed primary CNS tumors, with a focus on diffuse gliomas of grades II, III and IV, meningiomas from patients who are candidates for pharmacotherapy, and rare CNS tumors;
* Availability of adequate Human Biological Material (HBM): FFPE tissue sample from the primary and/or recurrent tumor and/or metastasis, obtained at the time of surgery or biopsy; minimal amount requested is detailed in the HBM guidelines. Inclusion of samples taken at any recurrence diagnosed during follow-up is strongly encouraged but optional;
* At least three months life expectancy;
* Written informed consent according to ICH/GCP and national/local regulations;
* Absence of exclusion criteria, such as active hepatitis B/C or HIV, second malignancies, severe organ dysfunction, or other comorbidities that will prevent inclusion into clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically confirmed brain cancer at any stage.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with brain malignancy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, MD, Study Chair — UniversitaetsSpital Zurich - Department of Neurology, Zurich, Switzerland
Locations (2):
- France (2):
  - CHRU de Lille, Lille
  - Assistance Publique - Hopitaux de Paris - La Pitie Salpetriere, Paris